CLINICAL TRIAL: NCT06818331
Title: Evaluation of Clinical Efficacy and Safety of Specific Mode Electroacupuncture Stimulation for Paclitaxel Across BBB Delivery in Patients With Postoperative Recurrence of Malignant Glioma: A Single-arm Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Xianming Lin, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSLL-KY-2024-079-01
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Glioma
Keywords: glioma; Specific Mode Electroacupuncture Stimulation; Paclitaxel; blood-brain barrier
MeSH Terms: conditions — Glioma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Patients in the treatment group received both paclitaxel(PTX) and a specific mode electroacupuncture stimulation（SMES） .
  Drug: Paclitaxel is administered intravenously at a dose of 135-175mg/m², repeated every 3 weeks.
  Device: SMES immediately after the ABX intravenous infusion began, the patient was placed in a supine position, the skin was routinely disinfected with 75% ethanol, and a stainless steel needle was inserted into GV20 and GV26.Then, the needles are stimulated by using an acupuncture point nerve stimulator with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off).
  Interventions: Other: SMES+PTX; Drug: Paclitaxel; Device: Specific mode electroacupuncture stimulation

INTERVENTIONS:
Other: SMES+PTX — This intervention involves the combined use of medication and device, where the specific mode electroacupuncture stimulation (SMES) intervention is administered simultaneously with the intravenous infusion of paclitaxel.
Drug: Paclitaxel — Paclitaxel is administered intravenously at a dose of 135-175mg/m², repeated every 3 weeks.
Device: Specific mode electroacupuncture stimulation — Patients assume a supine position. After routine skin disinfection with 75% ethanol, a stainless steel needle (size 0.25mm×40mm) is inserted into GV20 (Baihui), and another stainless steel needle (size 0.25mm×25mm, as described above) is inserted into GV26 (Shuigou). The acupoints are manually stimulated until the patient experiences soreness, distension, or heaviness (the "De Qi" response). Subsequently, the needles are stimulated using an acupuncture point nerve stimulator (HANS-200, Nanjing Jinsheng Ltd., China) at a frequency of 2/100 Hz and an intensity of 3 mA for 40 minutes (a homemade relay cycled power supply to the electrode, with 6 seconds on and 6 seconds off). The intervention is administered every three weeks, concurrently with paclitaxel treatment

SUMMARY:
Gliomas are the most common type of primary brain tumors, with the main treatment modalities including surgery, radiotherapy, and chemotherapy. However, gliomas are highly prone to recurrence, posing significant treatment challenges, especially for high-grade gliomas, which have a 5-year survival rate of only 5.5%. Paclitaxel (PTX) is a common chemotherapeutic agent, and its in vitro antitumor efficacy is 1400 times stronger than that of temozolomide (the first-line chemotherapy drug for gliomas). However, due to its large molecular weight (approximately 893 Da), it cannot cross the blood-brain barrier (BBB), preventing its use as a first-line treatment for gliomas. Preliminary research by our team has demonstrated that Specific Mode Electroacupuncture Stimulation (SMES) can open the BBB, increasing the concentration of PTX in tumor tissues, peritumoral tissues, and surrounding invasive tissues, thereby exerting antitumor effects. Therefore, this study aims to preliminarily observe the safety and efficacy of SMES combined with PTX in treating patients with postoperative recurrent high-grade gliomas.

ELIGIBILITY:
Inclusion criteria

1. WHO grade IV glioma as defined in the "Integrated Diagnosis and Treatment Guidelines for Glioma of the Chinese Anti-Cancer Association" (V2.0_2025 (20250110)).
2. Recurrence confirmed by cranial MRI after surgical resection.
3. According to the Response Assessment in Neuro-Oncology Criteria, version 2.0 (RANO 2.0) standards, there is at least one measurable lesion.
4. Age ≥ 18 years and ≤ 70 years, gender not limited.
5. If dexamethasone is used due to the space-occupying effect, the stable daily dose within 7 days before enrollment should be < 6 mg; if the dose of dexamethasone is being reduced, the average daily dose within 7 days before enrollment should be < 6 mg. Patients receiving dexamethasone treatment for reasons other than the space-occupying effect can still be enrolled.
6. Karnofsky Performance Status Score (KPS) ≥ 40 points or World Health Organization (WHO) Performance Status Score ≤ 3 points.
7. Good bone marrow function, liver and kidney function (within 14 days before treatment): a. Hemoglobin ≥ 90.0 g/L; b. White blood cells ≥ 3.0*10^9/L; c. Absolute neutrophil count ≥ 1500/µL (white blood cell count * neutrophil percentage); d. Platelets ≥ 100*10^9/µl; e. Total bilirubin (TbIL) ≤ 5.0 x ULN; f. Serum aspartate aminotransferase (SGOT) ≤ 3 x ULN and TbIL ≤ 3.0 x ULN; g. Creatinine ≤ 1.5 mg/dL, estimated glomerular filtration rate ≥ 30 mL/min to < 90 mL/min)
8. Able to receive electroacupuncture treatment and have good compliance.
9. Clear consciousness, pain perception and discrimination ability, and basic communication ability.
10. Signed the informed consent form and voluntarily participated in this study.

Exclusion criteria

1. Seizure attack, uncontrollable.
2. Those who are currently participating in other clinical trials or have completed other clinical trials within less than one month.
3. Those who have received treatment containing paclitaxel or similar drugs.
4. Those who have a severe allergy to paclitaxel or similar substances.
5. Pregnant or lactating women.
6. Those with diseases affecting cognitive function such as congenital dementia, or alcoholics, drug addicts or those with abuse of psychotropic substances.
7. Those with infected skin at the acupuncture site.
8. Patients with metallic foreign bodies in their bodies.
9. Those who cannot undergo cranial enhanced MRI examination.
10. Other acute or chronic diseases, mental disorders or abnormal laboratory test values that may increase the risk associated with participating in the study or the administration of the study drug, or interfere with the interpretation of study results, and the investigator determines that the patient does not meet the eligibility criteria for participation in the study.
11. Those who are undergoing other types of anti-tumor treatments simultaneously during the trial, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-02-24 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
4-month progression-free survival rate | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18.
  Comprehensive neurological examinations and MRI scans were performed at baseline to establish the initial disease status. These assessments were repeated at specified post-treatment time points (weeks 3, 6, 9, 12, 15, and 18) to evaluate changes compared to baseline. Responses, including complete response , partial response, stable disease , and progressive disease, were assessed according to the specific criteria outlined in the RANO 2.0 guidelines.Finally, the proportion of subjects in the intent-to-treat population with progression-free survival exceeding 4 months was calculated.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18.
  The questionnaire consists of 30 items and covers multiple dimensions, such as physical function, role function, emotional function, social function, quality of life, fatigue, pain, and other cancer-related symptoms.
The Neurological Assessment for Neuro-Oncology (NANO) | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18.
  NANO Scale quantitatively assesses nine neurological functions in patients, including gait, muscle strength, sensation, visual fields, facial strength, speech, cognition, and limb coordination, with each category scored between 0 to 3 or 0 to 2.
Overall survival(OS) | On the last day of weeks 3, 6, 9, 12, 15, and 18 during the treatment period; and then monthly during the follow-up phase for a total of 12 times.
  The time from enrollment to death for any reason (for lost-to-follow-up patients, the time of the last follow-up; for patients still alive at the end of the study, the time of the last follow-up).
Disease control rate | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18.
  Disease control rate refers to the proportion of patients in the intent-to-treat population who achieved complete response , partial response , or stable disease , as assessed by the RANO 2.0 criteria.
Objective response rate | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18.
  Objective response rate refers to the proportion of patients in the intent-to-treat population who achieved complete response or partial response , as assessed per the RANO 2.0 criteria.
Progression-free survival | On the last day of weeks 3, 6, 9, 12, 15, and 18 during the treatment period; and then monthly during the follow-up phase for a total of 12 times.
  Progression-free survival was defined as the time interval from the initiation of SMES combined with ABX treatment until the first occurrence of any of the following events: radiographic disease progression as determined by Response Assessment in Neuro-Oncology (RANO) version 2.0 criteria, the development of intolerable treatment-related adverse events leading to treatment discontinuation, or death due to any cause.
Duration of response | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18
  Duration of response was defined as the time interval between the first administration of SMES plus ABX therapy and the occurrence of disease progression.
Duration of Disease Control | baseline and 1-2 days before the end of weeks 3, 6, 9, 12, 15, and 18
  Duration of Disease Control was defined as the time interval from when a patient first achieved disease control (complete response , partial response , or stable disease until disease progression or death, whichever occurred first.
Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | On the 7th, 14th and 21st days of the 1st to 6th treatment cycles, each treatment cycle lasts for 21 days.
  Adverse reactions were recorded from the time of informed consent signing through the final visit, including any emerging symptoms, signs, and laboratory abnormalities. Common adverse reactions may include skin discomfort, pruritus, pain, etc., with severity graded into 5 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, China, Hangzhou City, Zhejiang Province, China

IPD SHARING:
Plan to Share IPD: No
The data and results of this study need to be confirmed by Lin Xianming

REFERENCES:
- [Background] Chamberlain MC, Kormanik P. Salvage chemotherapy with paclitaxel for recurrent primary brain tumors. J Clin Oncol. 1995 Aug;13(8):2066-71. doi: 10.1200/JCO.1995.13.8.2066. PMID 7636549
- [Background] Chang SM, Kuhn JG, Robins HI, Schold SC Jr, Spence AM, Berger MS, Mehta M, Pollack IF, Rankin C, Prados MD. A Phase II study of paclitaxel in patients with recurrent malignant glioma using different doses depending upon the concomitant use of anticonvulsants: a North American Brain Tumor Consortium report. Cancer. 2001 Jan 15;91(2):417-22. doi: 10.1002/1097-0142(20010115)91:23.0.co;2-9. PMID 11180089
- [Background] Barretina J, Caponigro G, Stransky N, Venkatesan K, Margolin AA, Kim S, Wilson CJ, Lehar J, Kryukov GV, Sonkin D, Reddy A, Liu M, Murray L, Berger MF, Monahan JE, Morais P, Meltzer J, Korejwa A, Jane-Valbuena J, Mapa FA, Thibault J, Bric-Furlong E, Raman P, Shipway A, Engels IH, Cheng J, Yu GK, Yu J, Aspesi P Jr, de Silva M, Jagtap K, Jones MD, Wang L, Hatton C, Palescandolo E, Gupta S, Mahan S, Sougnez C, Onofrio RC, Liefeld T, MacConaill L, Winckler W, Reich M, Li N, Mesirov JP, Gabriel SB, Getz G, Ardlie K, Chan V, Myer VE, Weber BL, Porter J, Warmuth M, Finan P, Harris JL, Meyerson M, Golub TR, Morrissey MP, Sellers WR, Schlegel R, Garraway LA. The Cancer Cell Line Encyclopedia enables predictive modelling of anticancer drug sensitivity. Nature. 2012 Mar 28;483(7391):603-7. doi: 10.1038/nature11003. PMID 22460905
- [Background] Caffery B, Lee JS, Alexander-Bryant AA. Vectors for Glioblastoma Gene Therapy: Viral & Non-Viral Delivery Strategies. Nanomaterials (Basel). 2019 Jan 16;9(1):105. doi: 10.3390/nano9010105. PMID 30654536
- [Background] Zhang S, Gong P, Zhang J, Mao X, Zhao Y, Wang H, Gan L, Lin X. Specific Frequency Electroacupuncture Stimulation Transiently Enhances the Permeability of the Blood-Brain Barrier and Induces Tight Junction Changes. Front Neurosci. 2020 Oct 6;14:582324. doi: 10.3389/fnins.2020.582324. eCollection 2020. PMID 33122995
- [Background] Park J, Aryal M, Vykhodtseva N, Zhang YZ, McDannold N. Evaluation of permeability, doxorubicin delivery, and drug retention in a rat brain tumor model after ultrasound-induced blood-tumor barrier disruption. J Control Release. 2017 Mar 28;250:77-85. doi: 10.1016/j.jconrel.2016.10.011. Epub 2016 Oct 11. PMID 27742444
- [Background] Siegal T, Rubinstein R, Bokstein F, Schwartz A, Lossos A, Shalom E, Chisin R, Gomori JM. In vivo assessment of the window of barrier opening after osmotic blood-brain barrier disruption in humans. J Neurosurg. 2000 Apr;92(4):599-605. doi: 10.3171/jns.2000.92.4.0599. PMID 10761648
- [Background] Graham-Gurysh EG, Murthy AB, Moore KM, Hingtgen SD, Bachelder EM, Ainslie KM. Synergistic drug combinations for a precision medicine approach to interstitial glioblastoma therapy. J Control Release. 2020 Jul 10;323:282-292. doi: 10.1016/j.jconrel.2020.04.028. Epub 2020 Apr 23. PMID 32335153
- [Background] Tosi U, Kommidi H, Adeuyan O, Guo H, Maachani UB, Chen N, Su T, Zhang G, Pisapia DJ, Dahmane N, Ting R, Souweidane MM. PET, image-guided HDAC inhibition of pediatric diffuse midline glioma improves survival in murine models. Sci Adv. 2020 Jul 24;6(30):eabb4105. doi: 10.1126/sciadv.abb4105. eCollection 2020 Jul. PMID 32832670
- [Background] Zagouri F, Zoumpourlis P, Le Rhun E, Bartsch R, Zografos E, Apostolidou K, Dimopoulos MA, Preusser M. Intrathecal administration of anti-HER2 treatment for the treatment of meningeal carcinomatosis in breast cancer: A metanalysis with meta-regression. Cancer Treat Rev. 2020 Aug;88:102046. doi: 10.1016/j.ctrv.2020.102046. Epub 2020 Jun 3. PMID 32599393
- [Background] Malani R, Fleisher M, Kumthekar P, Lin X, Omuro A, Groves MD, Lin NU, Melisko M, Lassman AB, Jeyapalan S, Seidman A, Skakodub A, Boire A, DeAngelis LM, Rosenblum M, Raizer J, Pentsova E. Cerebrospinal fluid circulating tumor cells as a quantifiable measurement of leptomeningeal metastases in patients with HER2 positive cancer. J Neurooncol. 2020 Jul;148(3):599-606. doi: 10.1007/s11060-020-03555-z. Epub 2020 Jun 6. PMID 32506369
- [Background] Fowler MJ, Cotter JD, Knight BE, Sevick-Muraca EM, Sandberg DI, Sirianni RW. Intrathecal drug delivery in the era of nanomedicine. Adv Drug Deliv Rev. 2020;165-166:77-95. doi: 10.1016/j.addr.2020.02.006. Epub 2020 Mar 3. PMID 32142739
- [Background] Agarwal S, Sane R, Oberoi R, Ohlfest JR, Elmquist WF. Delivery of molecularly targeted therapy to malignant glioma, a disease of the whole brain. Expert Rev Mol Med. 2011 May 13;13:e17. doi: 10.1017/S1462399411001888. PMID 21676290
- [Background] Cardoso FL, Brites D, Brito MA. Looking at the blood-brain barrier: molecular anatomy and possible investigation approaches. Brain Res Rev. 2010 Sep 24;64(2):328-63. doi: 10.1016/j.brainresrev.2010.05.003. Epub 2010 May 26. PMID 20685221
- [Background] Terstappen GC, Meyer AH, Bell RD, Zhang W. Strategies for delivering therapeutics across the blood-brain barrier. Nat Rev Drug Discov. 2021 May;20(5):362-383. doi: 10.1038/s41573-021-00139-y. Epub 2021 Mar 1. PMID 33649582
- [Background] Aldape K, Brindle KM, Chesler L, Chopra R, Gajjar A, Gilbert MR, Gottardo N, Gutmann DH, Hargrave D, Holland EC, Jones DTW, Joyce JA, Kearns P, Kieran MW, Mellinghoff IK, Merchant M, Pfister SM, Pollard SM, Ramaswamy V, Rich JN, Robinson GW, Rowitch DH, Sampson JH, Taylor MD, Workman P, Gilbertson RJ. Challenges to curing primary brain tumours. Nat Rev Clin Oncol. 2019 Aug;16(8):509-520. doi: 10.1038/s41571-019-0177-5. PMID 30733593
- [Background] Dmello C, Sonabend A, Arrieta VA, Zhang DY, Kanojia D, Chen L, Gould A, Zhang J, Kang SJ, Winter J, Horbinski C, Amidei C, Gyorffy B, Cordero A, Chang CL, Castro B, Hsu P, Ahmed AU, Lesniak MS, Stupp R, Sonabend AM. Translocon-associated Protein Subunit SSR3 Determines and Predicts Susceptibility to Paclitaxel in Breast Cancer and Glioblastoma. Clin Cancer Res. 2022 Jul 15;28(14):3156-3169. doi: 10.1158/1078-0432.CCR-21-2563. PMID 35552677
- [Background] Wick W, Stupp R, Beule AC, Bromberg J, Wick A, Ernemann U, Platten M, Marosi C, Mason WP, van den Bent M, Weller M, Rorden C, Karnath HO; European Organisation for Research and Treatment of Cancer and the National Cancer Institute of Canada Clinical Trials Group. A novel tool to analyze MRI recurrence patterns in glioblastoma. Neuro Oncol. 2008 Dec;10(6):1019-24. doi: 10.1215/15228517-2008-058. Epub 2008 Jul 31. PMID 18676355
- [Background] Rapp M, Baernreuther J, Turowski B, Steiger HJ, Sabel M, Kamp MA. Recurrence Pattern Analysis of Primary Glioblastoma. World Neurosurg. 2017 Jul;103:733-740. doi: 10.1016/j.wneu.2017.04.053. Epub 2017 Apr 19. PMID 28434963
- [Background] Weller M, Wick W, Aldape K, Brada M, Berger M, Pfister SM, Nishikawa R, Rosenthal M, Wen PY, Stupp R, Reifenberger G. Glioma. Nat Rev Dis Primers. 2015 Jul 16;1:15017. doi: 10.1038/nrdp.2015.17. PMID 27188790